CLINICAL TRIAL: NCT03922438
Title: Use of Cleft Margin Flap With Anterior Palatal Closure for Closure of Naso-alveolar Defect During Primary Cleft Lip Repair (Pilot Study).
Brief Title: Clinical Assessment of Usage of Cleft Margin Flap With Anterior Palatal Closure in Closure of Naso-alveolar Defect.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Yacoub Girgis, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CEBD-CU-2019-04-12
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Nasoalveolar Fistula (Defect)
Keywords: Cleft lip and palate; Cleft lip; Cleft alveolus; Cheiloplasty; Nasoalveolar fistula
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: Pilot study The eligible patients will be included in the study
Masking Description: No masking due to the nature of the intervention and the study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cleft margin flap with anterior palatal closure (Experimental): Usage of cleft margin flap with anterior palatal closure during primary cleft lip repair.
  Interventions: Procedure: usage of cleft margin flap with anterior palatal closure during primary cleft lip repair.

INTERVENTIONS:
Procedure: usage of cleft margin flap with anterior palatal closure during primary cleft lip repair. — Under general anesthesia, preparation of lip and palatal flaps will be done and then cleft margin flap which is designed to be inferiorly based will be used with anterior palatal closure in an attempt to decrease the incidence rate of naso-alveolar fistula (defect) that is usually occur and remain in those patients post-operatively.

SUMMARY:
During primary cleft lip repair in patients who were born with cleft lip and palate, usage of cleft margin flap with anterior palatal closure will be done in an attempt to close the Naso-alveolar fistula (defect) that usually occur and remain in those patients post-operatively.

DETAILED DESCRIPTION:
Cleft margin flap (that was discarded in the modified Millard's technique for cleft lip repair) with anterior palatal closure will be used during primary cleft lip repair in patients who were born with cleft lip and palate in an attempt to close the Naso-alveolar fistula (defect) that usually occur and remain in those patients post-operatively and this will be assessed in the predetermined follow up period.

Interventions:

General operative procedures

Eligible patients will be included in the study group:

* With the patient supine, general anesthesia will be induced, An uncuffed, oral, right angle endotracheal tube (RAE) will be placed and taped in the midline to the chin.
* The tube is further immobilized with a mouth pack.
* Head ring and shoulder rolls are placed. Sterile tapes will be placed over the closed eyelids. The face is prepared and draped.
* Reference points will be marked using brilliant green dye on a sharpened applicator stick.
* After careful marking, Approximately 3ml of 1% lidocaine with 1:200000 Epinephrines will be injected into the lip and alar base for homeostasis governed by heart rate of the patient.
* The lateral lip flap will first elevated with mucosal incision using number 15 blade scalpel at the gingivo-labial sulcus on the oral side and the release of the lateral lip segments will be achieved by dissecting over the lateral maxilla in the supra-periosteal plane.
* After this, a scalpel will be used to provide 1-2 mm of release of the skin from the underlying orbicularis oris muscle. This facilitates a 3 layer closure of mucosa, orbicularis oris muscle, and dermis. Then, the soft tissue attachments of the nasal base are separated from the piriform aperture. When the nasal dissection is complete, the surgeon is ready for closure of the lip deformity.
* Vomerine flap is done by doing incision on palatal side of the maxilla and vomer bone, then elevating mucoperiosteal flap on hard palate & undermining palatal mucosa.
* Closure of nasal lining.
* Mucosal flap obtained from part of the cleft near the lip was used as an inferior-based local flap. This flap was sutured to the anterior end of the mucoperiosteal flaps of the palate after it was passed from the alveolar cleft. The gingival mucosa on the alveolar cleft part was de-epithelialized, and lateral suturing of the flap was completed. In this way, not only the alveolar cleft but also the anterior palate cleft was corrected in this session.
* Skin hooks will be used to oppose the lip segments together to ensure that there is adequate release and minimal tension across the cleft wound. If too much tension exists, further dissection laterally or medially over the maxilla and superiorly along the bony piriform may be performed.
* Closure begins with 4-0 vicryl resorbable sutures placed in simple interrupted manner with the buried knots, to reconstituting the orbicularis oris muscular sphincter.

After this, the dermis will be closed by using 6-0 vicryl sutures. Approximation of the vermilion cutaneous borders must be precise, as any misalignment will become accentuated with subsequent growth.

5-0 vicryl sutures placed in the vermillion and the mucosa of the lip completing the closure.

Postoperative care:

* Cephalosporin antibiotic (Ceclor 125mg q12h) for five days.
* Otrivin saline nasal drops for 5 days.
* Mycostatin (Nystatin) Cream q8h for 5 days.
* Paracetamol drops 15ml.
* Fucidin cream ( sodium fusidate topical ) 3 times per day.
* Use of sterile tape as simple coverage for the wound for 5 days.
* Wash surgical wounds with soap & water until wound closes and heals.
* Massage the lip and columella with the cream downward with thumb once wound heals for 4-5 minutes twice a day for 3 months.

All patients will be evaluated at the following intervals:

* One week following Surgery
* One month following Surgery
* Six months following Surgery

ELIGIBILITY:
Inclusion Criteria:

* Non syndromic patients
* Medically fit for Surgery
* Patient with Primary, complete cleft lip
* Patient's age younger than six months

Exclusion Criteria:

* Patient with syndromic cleft lip
* Previous operated cases
* Incomplete cleft lip
* Patient older than six months
* Patients with any systemic condition

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Naso-alveolar fistula | 6 months postoperative.
  Naso-alveolar fistula will be assessed initially in the outpatient clinic by clinical examination and finally it will be re-assessed by usage of Methylene blue dye at time of cleft palate repair to assess the presence of any fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Beheiri, PhD, Study Director — Faculty of Oral and Dental Medicine- Cairo University; Mamdouh A AboulHassan, PhD, Study Director — Cairo University; Khaled A Salah Eldein, PhD, Study Director — Faculty of Oral and Dental Medicine- Cairo University; Sherif A Hassan, PhD, Study Director — Faculty of Oral and Dental Medicine- Cairo University; Dina Y Girgis, B.D.S, Principal Investigator — Faculty of Oral and Dental Medicine- Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcusson A, Akerlind I, Paulin G. Quality of life in adults with repaired complete cleft lip and palate. Cleft Palate Craniofac J. 2001 Jul;38(4):379-85. doi: 10.1597/1545-1569_2001_038_0379_qoliaw_2.0.co_2. PMID 11420018
- [Background] Mossey P. Epidemiology underpinning research in the aetiology of orofacial clefts. Orthod Craniofac Res. 2007 Aug;10(3):114-20. doi: 10.1111/j.1601-6343.2007.00398.x. PMID 17651127
- [Background] Mossey PA, Modell B. Epidemiology of oral clefts 2012: an international perspective. Front Oral Biol. 2012;16:1-18. doi: 10.1159/000337464. Epub 2012 Jun 25. PMID 22759666
- [Background] Wehby GL, Cassell CH. The impact of orofacial clefts on quality of life and healthcare use and costs. Oral Dis. 2010 Jan;16(1):3-10. doi: 10.1111/j.1601-0825.2009.01588.x. Epub 2009 Jul 27. PMID 19656316
- [Background] Wilhelmsen HR, Musgrave RH. Complications of cleft lip surgery. Cleft Palate J. 1966 Jul;3:223-31. No abstract available. PMID 5220833
- [Background] Kuna SK, Srinath N, Naveen BS, Hasan K. Comparison of Outcome of Modified Millard's Incision and Delaire's Functional Method in Primary Repair of Unilateral Cleft Lip: A Prospective Study. J Maxillofac Oral Surg. 2016 Jun;15(2):221-8. doi: 10.1007/s12663-015-0816-z. Epub 2015 Jul 25. PMID 27298546
- [Background] Isik D, Atik B, Tan O, Aktar S, Dogan M, Goktas U. Primary repair of the alveolar cleft. J Craniofac Surg. 2011 Nov;22(6):2224-6. doi: 10.1097/SCS.0b013e31823200c3. PMID 22075837
- [Background] Park YW, Kwon KJ, Kim MK. Double-layered reconstruction of the nasal floor in complete cleft deformity of the primary palate using superfluous lip tissue. Maxillofac Plast Reconstr Surg. 2015 Oct 13;37(1):35. doi: 10.1186/s40902-015-0035-z. eCollection 2015 Dec. PMID 26491651
- See also: Quality of life in adults with repaired complete cleft lip and palate — http://www.ncbi.nlm.nih.gov/pubmed/11420018
- See also: Epidemiology underpinning research in the aetiology of orofacial clefts — http://www.ncbi.nlm.nih.gov/pubmed/17651127
- See also: Epidemiology of oral clefts 2012: an international perspective — http://www.ncbi.nlm.nih.gov/pubmed/22759666
- See also: The Impact of Orofacial Clefts on Quality of Life and Health Care Use and Costs — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2905869/
- See also: Complications of cleft lip surgery. — http://www.ncbi.nlm.nih.gov/pubmed/5220833
- See also: Primary repair of the alveolar cleft — http://www.ncbi.nlm.nih.gov/pubmed/22075837
- See also: Double-layered reconstruction of the nasal floor in complete cleft deformity of the primary palate using superfluous lip tissue — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4604496/